CLINICAL TRIAL: NCT03224390
Title: A Pilot Study to Estimate the Impact of a Screening and Referral Service on Contraceptive Use
Acronym: E0108
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Moi University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2017-0406
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Results first posted 2019-07-19 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Contraception Behavior
Keywords: Contraception; Family Planning; Digital Health; Kenya; Unmet Need
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: The service (intervention) is available to anyone living in the catchment area, so it is not possible to randomly assign access to the service and estimate impact through a traditional randomized controlled trial (RCT). Likewise, at this early stage it is not be feasible to randomize access at a higher level, such as counties or subcounties. In situations like this, a variation on the traditional randomized controlled trial called a randomized encouragement design can be very effective.
  In a randomized encouragement design (RED), participants are randomized to receive an invitation or special encouragement to receive a treatment. Not everyone who is encouraged will take up the service, but as long as those randomly selected to receive the encouragement (the treatment group) use the service at a higher rate than the control group, the impact of the service can be estimated.
  For more details, see http://bit.ly/RED17protocol (linked in this record).
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Encouragement Arm (Experimental): Women randomized to the encouragement arm will receive an invitation via SMS to try the new digital family planning screening and referral service.
  Interventions: Other: digital family planning screening and referral service
- Control Arm (No Intervention): Women randomized to the control arm will receive a different set of SMS messages that do NOT include a special encouragement try the new digital family planning screening and referral service.

INTERVENTIONS:
Other: digital family planning screening and referral service — Clients text the service and receive a free call back to complete an automated family planning counseling session that results in a set of recommended methods that fit the client's preferences. The client is matched to family planning providers that offer these methods, and the service sends a referral code that the client can redeem at a facility. When someone receives a referral code, the service tracks them through their encounter with a provider to learn about their experience with the service, the provider, and their choice in contraception. The service also follows-up with clients who do not act on referrals to better understand their reasons and tries different behavioral nudges to promote uptake of contraception. The service does not pay costs the client may incur at a facility.
  Arms: Encouragement Arm

SUMMARY:
The specific aim of this pilot study is to estimate the impact of a new digital health service on the uptake of family planning among Kenyan women with an unmet need for contraception. Enrolled women will be randomized to a control arm or an encouragement arm that will receive a special invitation to try the new service.

DETAILED DESCRIPTION:
Based on global projections, meeting the unmet demand for contraceptives would prevent more than two-thirds of unintended pregnancies and more than two-thirds of maternal deaths. Voluntary family planning has also been shown to improve newborn health outcomes, advance women's empowerment, and bring socioeconomic benefits through reductions in fertility and population growth. Yet among the populations that would benefit the most from family planning, uptake remains too low.

The specific aim of this pilot study is to estimate the impact of a new digital health service on the uptake of family planning among Kenyan women with an unmet need for contraception. This service promotes uptake by offering free screening and referral. Women text the service for free, complete a short automated screening over the phone, and receive a list of recommended methods and a referral to local family planning providers offering those methods. The main hypothesis is that the service will increase the uptake of family planning among these users.

ELIGIBILITY:
Inclusion Criteria:

1. be between the ages of 18 and 35 (inclusive);
2. have an unmet need for family planning;
3. live in the service catchment area;
4. demonstrate phone ownership;
5. opt-in to receiving calls and/or SMS messages from the study team;
6. demonstrate basic ability to operate study tablet; and
7. consent to participate in the study.

Exclusion Criteria:

1. outside of the age range;
2. no unmet need for family planning;
3. live outside the service catchment area;
4. not able to demonstrate ownership of basic phone capable of receiving/making phone calls and receiving/sending SMS messages;
5. does not agree to receive calls and/or SMS messages from the study team;
6. does not demonstrate basic ability to operate study tablet; or
7. does not consent to participate in the study
8. not pregnant or <4 months postpartum

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Green, PhD, Principal Investigator — Duke University
Locations (1):
- Bungoma County, Bungoma, Kenya

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Green EP, Augustine A, Naanyu V, Hess AK, Kiwinda L. Developing a Digital Marketplace for Family Planning: Pilot Randomized Encouragement Trial. J Med Internet Res. 2018 Jul 31;20(7):e10756. doi: 10.2196/10756. PMID 30064968
- See also: Research design and analysis protocol — http://bit.ly/RED17protocol
- See also: Green et al. (2018). Developing a digital marketplace for family planning: Pilot randomized encouragement trial. Journal of Medical Internet Research, 20(7), e10756. — http://dx.doi.org/10.2196/10756

RESULTS

PARTICIPANT FLOW:
Groups:
- Encouragement Arm: One month after the end of the recruitment period, on October 2, 2017, women randomized to the encouragement arm received an invitation via SMS text message to try the service and complete a free family planning screening (plus bonus phone credit of approximately US $2, not conditional on the use of service).
- Control Arm: Women randomized to the control arm received a different set of messages thanking them for participating in the study; the control messages did not mention the investigational service.
Period: Overall Study
Arm/Group | Encouragement Arm | Control Arm
Started | 56 | 56
Completed | 29 | 21
Not Completed | 27 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Encouragement Arm | Control Arm | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (4.6) | 24.6 (5.0) | 24.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 112
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Luhya Tribe | 42 | 44 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Report Starting Any Modern Method of Contraception Since the Start of the Study
Description: Woman reports starting any modern method of contraception since the start of the study
Time Frame: 4-months post-encouragement
Measure: Count of Participants; unit: Participants
Arm/Group | Encouragement Arm | Control Arm
Number analyzed (Participants) | 56 | 56
Participants | 17 | 9
Statistical Analysis 1: Comparison: Encouragement Arm vs Control Arm; Test type: Superiority; Instrumental variables estimate = .41, 95% CI 2-sided [-.03 to .85]

2. Secondary Outcome: Uptake of Long-acting Contraception
Description: Woman reports starting any long-acting method of contraception since the start of the study
Time Frame: 1-month post-encouragement
Population: data were not collected
Arm/Group | Encouragement Arm | Control Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Encouragement Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56

LIMITATIONS AND CAVEATS:
The main limitation of this study was attrition. While attrition was not significantly associated with treatment assignment, found and unfound participants at endline differed on a few baseline characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT03224390/Prot_SAP_000.pdf